CLINICAL TRIAL: NCT04147429
Title: Reach Out and Read From Cradle to Clinic: A Novel Reach Out and Read Intervention in the Newborn Nursery
Brief Title: Newborn Nursery Reach Out and Read
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00102414
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-02

CONDITIONS: Literacy
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Newborns randomized to the usual care group will receive standard education about safe sleep practices, measuring temperatures and newborn feeding needs. This information will be accompanied by printed instructions that will be added to the family's discharge instructions. This reflects current practice in the Duke Hospital Newborn Nursery.
- Intervention (Experimental): In addition to usual care, families randomized to the intervention group will receive an early literacy intervention, delivered by a trained research assistant. To ensure intervention and delivery fidelity, the PI will meet with research assistants at bi-weekly intervals to review procedures and perform structured observations of intervention delivery.
  Interventions: Behavioral: Early Literacy Intervention

INTERVENTIONS:
Behavioral: Early Literacy Intervention — Similar to the standard Reach out and Read model, parents will be given a high-contrast board book, Cluck and Moo, and education about the importance of and how to engage with newborns in early shared reading behaviors. This will include instructive information for families about using books to stimulate newborns through pictures and spoken words.
  Arms: Intervention

SUMMARY:
The purpose of this research study is to learn new things about how parents and others who care for babies think about sharing books with their baby and how they might respond to guidance from their doctors. The study involves participants filling out a survey with questions about a newborn baby and thoughts about the baby's development. The study should not take more than an hour and fifteen minutes during the delivery hospital stay and another 20 minutes at the baby's one month well child visit by phone or emailed survey link. Participants may also be interviewed and asked some questions about these topics. The conversation will be audio recorded, and should last no more than 30 minutes. The survey should take no more than 15 minutes to complete. The participant and their child will be randomized, like flipping a coin, to either receive the study intervention book, Cluck and Moo, along with standard or care or solely standard of care at your time of hospital discharge. The greatest risks to this study would be feeling uncomfortable about answering some of the questions and potential risk of loss of confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Child delivered at Duke Hospital Birthing Center
* Families who can read and write in English
* Families with children born at >36 weeks gestation
* Families who plan to continue primary pediatric care with Duke Children's Primary Care

Exclusion Criteria:

* Parent with severe medical or mental health condition limiting ability to attend appointments
* Newborn with severe medical condition
* Families who plan to move out of state in the next 6 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-04-18 (Actual); Study Completion 2020-04-18 (Actual)

PRIMARY OUTCOMES:
Program acceptability as measured by survey data | 1 month
  Survey data will be analyzed using grounded theory.
Program acceptability as measured by structured interviews | 1 month
  The structured interviews will be evaluated and themes and subthemes will be identified using NVivo software.
Program feasibility assessed by determining the cost of books required for the intervention | 1 month
Program feasibility assessed by the time required to complete enrollment | 1 month
Program feasibility assessed by the time required to complete the intervention | 1 month
Program feasibility assessed by the number of eligible families enrolled in the study. | 1 month
Program feasibility assessed by the percentage of families who are followed through to study completion | 1 month

SECONDARY OUTCOMES:
Family's home literacy environment as measured by the READ subscale of the StimQ2-Infant. | 1 month
  Age appropriate items will be pulled from the StimQ2-Infant READ subscale. The StimQ2-Infant READ subscale measures a family's shared reading behaviors in the home.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Erickson, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No